CLINICAL TRIAL: NCT04498455
Title: Study of a Prebiotic Supplement to Mitigate Excessive Weight Gain Among Physicians in Residency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Principal Investigator, Leigh Greathouse, Assistant Professor of Nutrition Sciences, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1255329-5
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Weight Gain Trajectory; Metabolic Syndrome
Keywords: Fiber; Microbiome; Metabolism
MeSH Terms: conditions — Body-Weight Trajectory; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial of a fiber supplement [Prebiotin] compared to placebo [maltodextrin]
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Prebiotin
- Prebiotin (Active Comparator): Dietary Supplement: Prebiotin (oligofructose enriched inulin)
  Interventions: Dietary Supplement: Prebiotin

INTERVENTIONS:
Dietary Supplement: Prebiotin — Fructo-oligosaccharide dietary supplement powder

SUMMARY:
A randomized placebo controlled trial to determine if increased dietary fiber will prevent weight gain, inhibit adiposity and reduce perceived stress levels in residents at the Waco Family Health Center as the result of changes in distal gut microbiota composition and function.

DETAILED DESCRIPTION:
This study will utilize a single blind, placebo controlled, parallel design to assess the effect of dietary fiber [Prebiotin] on the gut microbiome, perceived stress, anthropometric variables, and clinical biomarkers of metabolism. All participants in this study will be resident physicians at the Family Health Center in Waco, TX. This population was selected based on pilot data indicating they are at a greater risk for weight gain and have higher levels of stress than the average population. The goal is to recruit 40 participants for a 12 week intervention trial.

ELIGIBILITY:
Inclusion Criteria:

* Currently a resident in training at the Family Health Center in their first year.

Exclusion Criteria:

* Pregnancy
* Currently on prescribed metformin or NSAIDS
* A diagnosed gastro-intestinal disease (i.e. irritable bowel syndrome or Crohn's disease)
* Known allergy to the supplement, placebo, or provided meal replacements
* Antibiotic use within the last 3 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 12 weeks
  The investigators will use the following procedure to assess the effect of Prebiotin (OEI) on changes in body weight: there will be two test days: a) baseline (Day 0), prior to randomization to OEI or placebo; and b) week 12, following the 11 week course of OEI/placebo treatment. The investigators will use OEI for the inulin challenge. Change in body weight will be quantified by bio electrical impedance.

CONTACTS AND LOCATIONS:
Overall Officials: LesLee Funderburk, Ph.D., Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data

REFERENCES:
- See also: Study analysis — https://greathouselab.github.io/Fiber_Intervention_Study/